CLINICAL TRIAL: NCT03935776
Title: The Effect of Lifestyle and Risk Factor Modification on Occlusive Peripheral Arterial Disease Outcomes: Standard Healthcare vs Structured Programme
Brief Title: Lifestyle Modification Programme for Patients With Peripheral Arterial Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Vascular Institute, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WVI-PAD
Record Dates: First submitted 2019-02-15; First posted 2019-05-02 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Peripheral arterial disease; Risk factor modifications; Cardiovascular risk factors
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: This is a randomised, parallel group, active-control trial, with patients randomised in a 1:1 ratio
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of trial participants and care providers is not possible because of obvious differences between the interventions. However, the investigator, the outcomes assessor and statistician are blinded to treatment received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk Factors Modification Programme (Experimental): * Patients in the intervention arm will attend a 12-week intensive lifestyle programme.
  * The intervention includes weekly exercise class and educational workshops, serial blood pressure, body mass index, glucose and lipid measurements.
    * Weekly multidisciplinary team meetings and targeted and protocol pharmacotherapy to support lifestyle changes.
  Interventions: Behavioral: Risk Factors Modification Programme
- Standard Healthcare (Active Comparator): The control group will receive information and advice to the patients to modify their lifestyles but without providing a structured intervention or an individualised plan.
  Interventions: Behavioral: Standard Healthcare

INTERVENTIONS:
Behavioral: Risk Factors Modification Programme — 12- week supervised risk factor modification programme derived from the Euroaction study standards
  Arms: Risk Factors Modification Programme
Behavioral: Standard Healthcare — Patients are advised to adjust lifestyle without the support of the structured supervised programme
  Arms: Standard Healthcare

SUMMARY:
This trial randomises patients with occlusive peripheral arterial disease, to be managed either by providing a 12-week structured lifestyle modification programme, or standard healthcare.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects more than 200 million of the global population. PAD represents a marker for premature cardiovascular events.

Despite the high prevalence of PAD and the strong association with cardiovascular morbidity and mortality, patients with PAD are less likely to receive appropriate treatment for their atherosclerotic risk factors than those who are being treated for coronary artery disease.

Because PAD represents a peripheral manifestation of atherosclerosis, most traditional and novel cardiovascular risk factors are strongly associated with this condition. Smoking, diabetes, hyperlipidaemia, hypertension, unhealthy diet, and physical inactivity were identified as significant modifiable risk factors that should be targeted for secondary prevention.

Atherosclerotic risk factor identification and modification plays an important role in reducing the number of adverse outcomes among patients with atherosclerosis. Risk reduction therapy decreases the risk of cardiovascular mortality and morbidity in patients with PAD. Because of the efficacy of these techniques, several expert committees have recommended their use in patients with PAD. Despite clear guidelines, several studies have shown that patients with PAD are routinely undertreated for these risk factors, which may contribute to high rates of morbidity and mortality.

Our trial will evaluate the impact of a 12-week, structured lifestyle and risk factor modification programme on medical and lifestyle risk factors modification, as well as on clinical vascular outcomes, among patients with peripheral arterial disease. We will compare these outcomes to that of standard healthcare traditionally provided to this high-risk patient group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Provide written informed consent
* PAD: diagnosed by at least one of the following:

  * Ankle-brachial index of less than 0.90 in at least one lower extremity(10)
  * Toe brachial index of less than 0.609
  * Evidence of arterial occlusive disease in one lower extremity detected by duplex ultrasonography, computed tomographic angiography, or magnetic resonance angiography(10)
* Symptomatic PAD (Rutherford category 2 and above(11)
* Patients should have at least one of the following risk factors:
* Blood pressure > 140/80 mmHg
* Fasting Blood Sugar (FBS) >53 mmol/mol
* HbA1c >7%
* Total cholesterol >5 mmol/L
* LDL cholesterol >2.6 mmol/L
* Triglycerides >1.7 mmol/L
* HDL <1.0 mmol/L in men and <1.2 mmol/L in women
* Physical activity less 30 minutes for 5 days per week
* BMI 25>kg/m2
* Waist circumference >80 cm in women, and >94 cm in men.
* Current smoker or exposure to tobacco in any form
* Unhealthy diet, Mediterranean diet score less than 10 points

Exclusion Criteria:

* Rutherford category zero or one(11)
* Involvement in another clinical trial in the previous six months
* Legal incapacity
* Inadequate English language
* Significant cognitive impairment or mental illness
* Inadequate English language
* Significant cognitive impairment or mental illness
* Refusal to participate in a certain part of the intervention
* Mental and physical inability to participate in the structured programme
* Pregnant (confirmed by β-human chorionic gonadotropion (HCG) analysis).
* Contraindication to anticoagulation and antiplatelet medications or any of the risk factors treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Lifestyle and medical risk factor modification | at 12 weeks
  Achieving target Improvement in lifestyle risk factors. Target improvement will be considered if the patient achieves any one or more of the following:
  1. Smoking cessation
  2. Body mass index 20-25 (kg/m^2). BMI is calculated by dividing body weight in kilograms by the square of height in meters
  3. Glycosylated haemoglobin (HbA1c) less than 7%
  4. Total Cholesterol less than 5.0 mmol/L

SECONDARY OUTCOMES:
Amputation free survival | 1 year
  if the patient underwent a major amputation and level of amputation
Re-intervention or stenosis rate | 1 year
  Any re-intervention or stenosis among patients who already underwent vascular surgery
Freedom from major adverse cardiovascular events (MACE) and major adverse limb events (MALE) | 1 year
  If the patient developed a major adverse cardiovascular event (MACE) or major adverse limb event (MALE)
Revascularisation-free survival | 1 year
  if the patient underwent any revascularisation procedure
Health related quality of life | 1 year
  assessed using the Dartmouth Cooperative Information Project (COOP) charts at enrolment and after one year.
  The COOP charts measure six core aspects of functional status: physical fitness, feelings, daily activities, social activities, change in health, pain, and overall health. The instrument consists of six charts, referring to the above mentioned aspects of functioning. Each chart consists of a simple title, a question referring to the status of the patient and an ordinal five-point response scale illustrated with a simple drawing.
  Each item is rated on this five-point ordinal scale ranging from 1 (no limitation at all) to 5 (severely limited); for 'change in health' score 1 means 'much better' and score 5 'much worse'. The designers do not advocate summing the responses to gain a single index ﬁgure of health status.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Tawfick, MB BcH,MRCSI, Principal Investigator — Western Vascular Institute, Ireland; Sherif Sultan, MB BcH,MRCSI, Principal Investigator — Western Vascular Institute, Ireland; Marah Elfghi, MB BcH, MSc, Study Director — Western Vascular Institute, Ireland
Locations (1):
- Department of Vascular Surgery, Western Vascular Institute, Galway University Hospital, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data of primary and secondary outcomes, could be made available to other researchers by request, while maintaining participant confidentiality

REFERENCES:
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Newman AB, Shemanski L, Manolio TA, Cushman M, Mittelmark M, Polak JF, Powe NR, Siscovick D. Ankle-arm index as a predictor of cardiovascular disease and mortality in the Cardiovascular Health Study. The Cardiovascular Health Study Group. Arterioscler Thromb Vasc Biol. 1999 Mar;19(3):538-45. doi: 10.1161/01.atv.19.3.538. PMID 10073955
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Becker GJ, McClenny TE, Kovacs ME, Raabe RD, Katzen BT. The importance of increasing public and physician awareness of peripheral arterial disease. J Vasc Interv Radiol. 2002 Jan;13(1):7-11. doi: 10.1016/s1051-0443(07)60002-5. No abstract available. PMID 11788688
- [Background] Criqui MH, Fronek A, Klauber MR, Barrett-Connor E, Gabriel S. The sensitivity, specificity, and predictive value of traditional clinical evaluation of peripheral arterial disease: results from noninvasive testing in a defined population. Circulation. 1985 Mar;71(3):516-22. doi: 10.1161/01.cir.71.3.516. PMID 3156007
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Background] Shen C, Li W. [Interpretation and consideration of the Society for Vascular Surgery practice guidelines for atherosclerotic occlusive disease of the lower extremities management of asymptomatic disease and claudication]. Zhonghua Wai Ke Za Zhi. 2016 Feb 1;54(2):81-3. doi: 10.3760/cma.j.issn.0529-5815.2016.02.001. Chinese. PMID 26876071
- [Background] Lu JT, Creager MA. The relationship of cigarette smoking to peripheral arterial disease. Rev Cardiovasc Med. 2004 Fall;5(4):189-93. PMID 15580157
- [Background] Mahe G, Kaladji A, Le Faucheur A, Jaquinandi V. Internal Iliac Artery Disease Management: Still Absent in the Update to TASC II (Inter-Society Consensus for the Management of Peripheral Arterial Disease). J Endovasc Ther. 2016 Feb;23(1):233-4. doi: 10.1177/1526602815621757. No abstract available. PMID 26763263
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Derived] Elfghi M, Jordan F, Dunne D, Gibson I, Jones J, Flaherty G, Sultan S, Tawfick W. The effect of lifestyle and risk factor modification on occlusive peripheral arterial disease outcomes: standard healthcare vs structured programme-for a randomised controlled trial protocol. Trials. 2021 Feb 13;22(1):138. doi: 10.1186/s13063-021-05087-x. PMID 33581715